CLINICAL TRIAL: NCT01651624
Title: Comparison Between Faecal Occult Blood Test (FOBT), Computed Tomographic Colonography (CTC) With Computer Aided Diagnosis (CAD) and Colonoscopy as a Primary Screening Test for Colorectal Cancer. Validation of a Teleradiology Model. Biological Banking in Subjects Recruited for Colonoscopy or CTC.
Brief Title: Screening for Colorectal Cancer With FOBT, Virtual Colonoscopy and Optical Colonoscopy. A Randomized Clinical Trial in the Florence District
Acronym: SAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Prevention and Research Institute, Italy (Other)
Collaborators: University of Florence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: D65C09002710007; 432/10 (Other: Local Ethics Committee of Local Health Unit of Florence)
Record Dates: First submitted 2012-07-20; First posted 2012-07-27 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Screening; Fecal Occult Blood Test; CT Colonography; Virtual Colonoscopy; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Computed tomographic colonography (CTC), reduced prep (Experimental): Subjects invited to undergo CTC with reduced cathartic preparation
  Interventions: Other: Invitation to screening
- Computed tomographic colonography (CTC), standard prep (Experimental): Subjects invited to undergo CTC with standard bowel preparation
  Interventions: Other: Invitation to screening
- Faecal occult blood test (FOBT) (Active Comparator): Subjects invited to undergo FOBT
  Interventions: Other: Invitation to screening
- Colonoscopy (Experimental): Subjects invited to undergo colonoscopy
  Interventions: Other: Invitation to screening

INTERVENTIONS:
Other: Invitation to screening

SUMMARY:
RATIONALE: Computed tomographic colonography (CTC) has proven to be accurate in detecting colorectal neoplasms and may be a primary test in colorectal cancer screening.

PURPOSE: This clinical trial will compare participation rate, diagnostic yield and costs of computed tomographic colonography, faecal occult blood test (FOBT) and colonoscopy (CO) as a primary screening test in a population-based programme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary objectives:

* To compare the participation rate to faecal occult blood test (FOBT), computed tomographic colonography (CTC) and colonoscopy (CO) as a primary screening test in a population-based programme for colorectal cancer.
* To compare the participation rate to CTC with reduced cathartic preparation versus CTC with standard bowel preparation.
* To compare the detection rate for cancer or advanced adenomas of CTC with computer aided diagnosis (CAD) versus three rounds of FOBT every second year.
* To evaluate referral rate for colonoscopy induced by primary CTC versus three rounds of FOBT every second year.
* To compare costs of the three screening strategies.

Secondary objectives:

* To compare the expected and perceived discomfort of colonoscopy and computed tomographic colonography as assessed with a structured questionnaire.
* To evaluate the rate of complications in each group.
* To validate a teleradiology model for computed tomographic colonography.
* To create a biological bank of blood and stool specimens from subjects who undergo computed tomographic colonography, primary colonoscopy and second level colonoscopy.

DESIGN:

14,000 subjects aged 55-64 years, living in the Florence District and never screened for colorectal cancer, will be randomized in 3 arms:

* group 1 (5,000 persons) invited to CTC (divided into: subgroup 1A with reduced cathartic preparation and subgroup 1B with standard bowel preparation);
* group 2 (8,000 persons) invited to biannual FOBT for 3 rounds;
* group 3 (1,000 persons) invited to CO.

Subjects of each group will be invited by mail to undergo the selected test. Individuals of each group will receive an invitation letter and an information leaflet, containing information about colorectal cancer, importance of screening, and advantages and possible risks of the selected test.

Invitation letter for the FOBT group contains instructions on how to pick-up the kit test at the nearest pharmacy. The FOBT screening test adopted is OC-SENSOR DIANA (Eiken Chemical Co., Tokyo, Japan), a quantitative, completely automated immunochemical test, based on latex agglutination. Positivity threshold is set at 100 ng/ml of sample solution. Invited subjects are asked to collect a single sample of faeces, without dietary restrictions. Sample are retuned according to the routine procedure of Florence screening programme.

Invitation letter for CTC and colonoscopy contains a phone number and an email address of the screening centre. All invitees have the option to call or send an email to the screening centre in order to receive an appointment for a prior consultation. All non-responders will receive a remainder by mail after three months. Non-responders to reminder will be invited to FOBT according with current screening procedure.

Subjects who accept invitation for CTC or CO will have a consultation at the screening centre with a trained nurse. During the consultation subjects will be informed about the study protocol, the screening examination to which they are invited, the bowel preparation, and the management in case of positive results. All subjects tested positive to FOBT or CTC (mass or at least one polyp ≥ 6 mm) will be invited to undergo total colonoscopy. Then, subjects will be scheduled for the selected examination (CTC or CO).

ELIGIBILITY:
Inclusion Criteria:

* Never invited to previous colorectal cancer screening.

Exclusion Criteria:

* Personal history of colorectal cancer or colonic advanced adenomas.
* Inflammatory bowel disease (IBD).
* Previous five years complete colonoscopy or previous two years faecal occult blood test (FOBT).

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16087 (Actual)
Dates: Start 2012-12; Primary Completion 2018-11-25 (Actual); Study Completion 2018-11-25 (Actual)

PRIMARY OUTCOMES:
Participation rate to faecal occult blood test (FOBT), computed tomographic colonography (CTC) and colonoscopy | 2 years
Detection rate for cancer or advanced adenomas of CTC versus three rounds of FOBT every second year | 6 years
Referral rate for colonoscopy induced by primary CTC versus three rounds of FOBT every second year | 6 years
Costs of the three different screening strategies proposed | 6 years

SECONDARY OUTCOMES:
Expected and perceived burden of colonoscopy and CTC | 2 years
Number and type of complications in all groups | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Milani, MD, Principal Investigator — University of Florence; Grazia Grazzini, MD, Study Director — Cancer Prevention and Research Institute, Italy
Locations (1):
- Cancer Prevention and Research Institute, ISPO, Florence, FI, Italy

REFERENCES:
- [Derived] Sali L, Ventura L, Mascalchi M, Falchini M, Mallardi B, Carozzi F, Milani S, Zappa M, Grazzini G, Mantellini P. Single CT colonography versus three rounds of faecal immunochemical test for population-based screening of colorectal cancer (SAVE): a randomised controlled trial. Lancet Gastroenterol Hepatol. 2022 Nov;7(11):1016-1023. doi: 10.1016/S2468-1253(22)00269-2. Epub 2022 Sep 16. PMID 36116454
- [Derived] Sali L, Grazzini G, Carozzi F, Castiglione G, Falchini M, Mallardi B, Mantellini P, Ventura L, Regge D, Zappa M, Mascalchi M, Milani S. Screening for colorectal cancer with FOBT, virtual colonoscopy and optical colonoscopy: study protocol for a randomized controlled trial in the Florence district (SAVE study). Trials. 2013 Mar 15;14:74. doi: 10.1186/1745-6215-14-74. PMID 23497601